CLINICAL TRIAL: NCT02048605
Title: Basel Training Study II: Training of Psychosocial Skills for Patients With Parkinson's Disease
Brief Title: Training of Psychosocial Skills Based on Cognitive Behavioural Therapy for Patients With Parkinson's Disease
Acronym: CBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Parkinson Schweiz (Other); Bangerter-Rhyner Foundation (Unknown); AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BSLTraining2
Record Dates: First submitted 2014-01-23; First posted 2014-01-29 (Estimated); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Parkinson's Disease; Mild Cognitive Impairment
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psycho-social (CBT) based training (Experimental): Psycho-social Training in Neurological Diseases - Parkinson's Disease ( Training according to Ellgring et al., 2006)
  Interventions: Behavioral: Psycho-social CBT based training
- Unspecific group training (Placebo Comparator): Health Enhancement Program
  The validation of an active control intervention for Mindfulness Based Stress Reduction (MBSR) (MacCoon et al., 2012)
  Interventions: Behavioral: Unspecific group training

INTERVENTIONS:
Behavioral: Psycho-social CBT based training — Number of Sessions: 9x Content: cognitive behavioral group-training-program to reduce stress and augment quality of life.
  Arms: Psycho-social (CBT) based training
Behavioral: Unspecific group training — Number of sessions: 9x Content: Music or Art Therapy Nutrition Education around Food Functional Movement Physical Activity Group discussion
  Other Names: Health Enhancement Program
  Arms: Unspecific group training

SUMMARY:
Patients with Parkinson's disease (PD) will be trained using a cognitive behavioral group-training-program to reduce stress and augment quality of life. An unspecific group with the same amount and frequency of meetings is used as a control group. For the evaluation of the training effects, scales to assess quality of life, analyses of psychopathological variations as well as neurocognitive tests will be used. Protocol amendment in 1-2017: addition of FU year 3 and year 5.

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic Parkinson's disease according to United Kingdom Parkinson's Disease Brain Bank Criteria, being either cognitively normal, suffering from Mild Cognitive Impairment or having mild dementia. Patients must be able to give their written informed consent.

Exclusion Criteria:

* Moderate or severe dementia (DMS-IV, Mini Mental Status (MMS) <24), other neurological or psychiatric diseases of the brain not related to PD, secondary parkinsonism, physical impairment hindering the adequate execution of the training, insufficient knowledge of German or pregnancy are exclusion criteria. Deep Brain Stimulation (DBS) is no exclusion criterion.

Ages: 45 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Schedule for the Evaluation of Individual Quality of Life-Direct Weighting (SeiQol-DW) | Before and after 9 weeks of training, After 6-month

SECONDARY OUTCOMES:
Scale for the assessment of management of daily living (Alltagsbewältigungsskala: A-B-S) | Before and after 9 weeks training, after 6 month

OTHER OUTCOMES:
Burden questionnaire for Patients with Parkinson's Disease (Belastungsfragebogen) | Before and after 9 weeks of training, after 6 month
  Questionnaire for measuring psychosocial problems, no official english translation available.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Fuhr, Prof., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Result] Hadinia A, Meyer A, Bruegger V, Hatz F, Nowak K, Taub E, Nyberg E, Stieglitz RD, Fuhr P, Gschwandtner U. Cognitive Behavioral Group Therapy Reduces Stress and Improves the Quality of Life in Patients with Parkinson's Disease. Front Psychol. 2017 Jan 4;7:1975. doi: 10.3389/fpsyg.2016.01975. eCollection 2016. PMID 28101066
- See also: Click here for more information about this study — http://parkinson-team.ch/